CLINICAL TRIAL: NCT03700307
Title: Changes in Left Atrial Function After Respective Treatments of Persistent Atrial Fibrillation With Circumferential Pulmonary Vein Isolation, Circumferential Pulmonary Vein and Left Atrial Linear Isolation Using Cryoballoon Ablation and Effects of the Application of Statin Drugs
Brief Title: Effects of Different Surgical Methods for Persistent Atrial Fibrillation Combined With the Application of Statin Drugs on Left Atrial Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Second Hospital of Hebei Medical University (Other)
Responsible Party: Principal Investigator, xieruiqin, director of cardiology department, The Second Hospital of Hebei Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: XieruiqindoctorAF
Record Dates: First submitted 2018-08-28; First posted 2018-10-09 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2020-03

CONDITIONS: Persistent Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- pulmonary vein isolation (Experimental): patients will receive circumferential pulmonary vein isolation using cryoballoon ablation
  Interventions: Procedure: Cryoballoon ablation
- pulmonary vein and left atrial roof linear isol (Experimental): patients will receive circumferential pulmonary vein and left atrial roof linear isolation using cryoballoon ablation
  Interventions: Procedure: Cryoballoon ablation

INTERVENTIONS:
Procedure: Cryoballoon ablation — Cryoablation is performed using a single cryoballoon.In general, the cryoablation of each pulmonary vein is carried out twice.

SUMMARY:
A total of 164 patients with persistent atrial fibrillation, who are planned to undergo treatment with cryoballoon ablation, will be randomly allocated into two groups. These patients will receive circumferential pulmonary vein isolation, circumferential pulmonary vein and left atrial roof linear isolation using cryoballoon ablation(allocation ratio, 1:1). Patients in each group will be randomly allocated into the statin treatment group and non-statin treatment group (allocation ratio, 1:1). Real-time 3D ultrasound and 2D ultrasound examinations and measurement of left atrial function are carried out for all patients before the operation, and at 1, 2, 3 and 4 weeks and 2, 3, 6, 9 and 12 months after the operation. Preoperative transesophageal echocardiography will be carried out in all patients to measure the left atrial appendage function. All ultrasound data will be stored and a professional director from the ultrasound room will be invited for quantitative analysis. Indicators for ultrasonography include: left atrial anterior and posterior diameter, left atrial volume, left atrial volume index, mitral e ", E peak, A peak, velocity time integral (VTI), left atrial ejection fraction, left atrial strain, strain rate and left atrial appendage emptying velocity. Blood samples are extracted in all patients to detect routine blood, troponin I, D-D dimer, oral anticoagulant monitoring and other biochemical parameters such as blood lipids before the operation and at 1, 2, 3 and 4 weeks and 1, 2 and 3 months after the operation. This study will clarify whether these different operation methods have different effects on the recovery of postoperative left atrial function in patients with persistent atrial fibrillation, and whether changes in left atrial function are related to indicators such as inflammation, blood clotting and myocardial injury. Furthermore, this study will investigate whether the application of statin drugs can improve postoperative left atrial function by affecting these indicators. In addition, the operation method has been improved targeting at the disadvantage of the greater amount of X-ray exposure during cryoballoon ablation for persistent atrial fibrillation. Circumferential pulmonary vein isolation is combined with left atrial roof linear isolation，and related indicators such as the success rate of the operation, intraoperative complications, postoperative recurrence rate and the amount of x-ray exposure are compared among two groups. At the same time, biochemical indicators of inflammation, blood clotting and myocardial injury such as blood routine, myocardial enzyme, troponin I and D-D dimmer are detected to analyze and determine which indicators are related to the postoperative recurrence of atrial fibrillation, the incidence of postoperative thrombosis and the recovery of postoperative left atrial function.

DETAILED DESCRIPTION:
A total of 164 patients with persistent atrial fibrillation(AF), who are planned to undergo treatment with cryoballoon ablation, will be randomly allocated into two groups.

1. Each patient randomly allocated into the circumferential pulmonary vein isolation group receives circumferential pulmonary vein isolation using cryoballoon ablation, and no additional isolation or ablation is performed in the extrapulmonary sites unless the patient is diagnosed with right atrial flutter before the operation.The investigators will carry out tricuspid isthmus ablation during the operation for patients with a preoperative diagnosis of right atrial flutter. All patients will undergo the remodeling of pulmonary vein-left atrium under CT before the operation to understand the structures of the left atrium and pulmonary veins. Patients who have recurrent atrial fibrillations within the first three months during postoperative follow-up will not be considered for repeated the operation.
2. Each patient randomly allocated into the circumferential pulmonary vein and left atrial linear isolation group receives circumferential pulmonary vein and left atrial roof linear isolation using cryoballoon ablation,no additional isolation or ablation is performed in the extra sites unless the patient is diagnosed with right atrial flutter before the operation. The investigators will carry out tricuspid isthmus ablation during the operation for patients with a preoperative diagnosis of right atrial flutter. All patients will undergo the remodeling of pulmonary vein-left atrium under CT before the operation to understand the structures of the left atrium and pulmonary veins. Patients who have recurrent atrial fibrillations within the first three months during postoperative follow-up will not be considered for repeated the operation. Cryoablation is performed using a single cryoballoon. The diameter of the cryoballoon (Arctic Front Advance™ Cardiac CryoAblation Catheter; Medtronic, Minneapolis, MN) is determined as 28 mm or 23 mm according to pulmonary venography results. After passing through the transseptal sheath, the cryoballoon catheter enters into the left atrium and is continuously infused with heparin saline through a 12 French(12F) oriented sheath. The circular mapping catheter (Achieve, Medtronic) will pass through the balloon catheter and first enter into the pulmonary vein lumen. It is placed as close as possible into the pulmonary vein to record original pulmonary vein potentials and carry out intraoperative real-time monitoring of the isolation of pulmonary vein potentials.

   The balloon is inflated at the entrance of the pulmonary vein. The mapping confirms that the balloon blocks the entrance of the pulmonary vein. After blocking of the entrance of the pulmonary vein is enhanced, liquid nitrogen is injected for cryoablation, which lasts for 240 seconds each time. Before performing right pulmonary vein ablation, a secondary catheter is placed into the superior vena cava during the cryoablation. A cycle length of 999 ms is taken to continuously make the right phrenic nerve pulsate. If diaphragm movement is weakened or disappears, the cryoablation will be immediately stopped. In general, the cryoablation of each pulmonary vein is carried out twice. If the cryoablation is unsuccessful for twice, an additional cryoablation can be carried out; but the number of times of pulmonary vein cryoablation should not be more than five.The patients randomly allocated into the circumferential pulmonary vein and left atrial linear isolation group receives circumferential pulmonary vein and left atrial roof linear isolation using cryoballoon ablation
3. Examinations of real-time 3D ultrasound, 2D ultrasound, transesophageal echocardiography and Doppler are carried out to measure the left atrial size and function for all patients before the operation and at 1, 2, 3 and 4 weeks and 2, 3, 6, 9 and 12 months after the operation (iE33 machines equipped with X3, Philips). Measurement of left atrial anterior and posterior diameter: the left ventricular long axis next to the sternum is taken to measure the left atrial anterior and posterior diameter in the end systolic period of the left atrium; mitral e ": apical four-chamber view, sampling volume locates in the site of the mitral annular septum, and early diastolic blood flow velocity is measured; E peak: mitral valve early diastolic flow velocity; A peak: mitral valve late diastolic flow velocity; mitral valve velocity time integral. Measurement of left atrial ejection fraction: Five references sites are taken in the atrium, including four reference sites located in the front, lower, lateral and septal side of the top of the atrium, and one reference site located at the level of the mitral annulus. During the cardiac cycle, volumes at three time points will be measured. ① LAMax means that the left atrial volume is measured in the end systolic period before the opening and closing of the mitral valve, ② LAMin means that the left atrial volume is measured at end diastolic period before the closing of the mitral valve, and ③ LApreA means that the left atrial volume is measured before the appearance of the corresponding body surface ECG P-wave. These are obtained through the following formulas using the surface area index and left atrial function: the left atrial ejection fraction (LAEF) = [(LAMax- LAMin) / LAMax] × 100% - the active atrial emptying rate; the active left atrial emptying rate (LAactive) = [(LApreA - LAmin ) / LApreA] × 100% - passive atrial emptying rate; the passive left atrial emptying rate (LA passive) = [(LAmax - LApreA) / LAmax] × 100% - the atrial expansion index. The left atrial strain (four chambers, two-chamber): three reference sites are placed using Qlab software (CMQ, Philips Medical Systems). In four-chamber view, three reference sites are respectively placed in the mitral annular septum, the free wall of the mitral annulus and the top of the atrium. In two-chamber view, three reference sites are respectively placed in the front wall of the atrium, the free wall of the mitral annulus and the top of the atrium. The software will automatically track atrial muscle movement and work out the left atrial strain and left atrial strain rate. All patients will undergo preoperative transesophageal echocardiography to obtain the left atrial appendage (LAA) emptying velocity.
4. Patients in the two groups of cryoballoon ablation, will be randomly allocated again into the statin treatment group and non-statin treatment group. Patients in the statin treatment group will orally receive 20 mg of atorvastatin per night (Pfizer) for three days before the operation and three months after the operation. Forms are filled in for all patients before the operation to record medical histories and related biochemical parameters in detail (including all blood routine indicators [Neutrophil%(NE%), Lymphocyte% (LY%), NE/LY], International Normalized Ratio (INR), enzymes, troponin, blood lipids and D-D dimer). The above-mentioned blood biochemical parameters are reexamined for all patients at 1, 2, 3 and 4 weeks and 1, 2 and 3 months after the operation. In addition to the above-described echocardiographic reexamination and blood samples, the content of the follow-up after ablation also includes symptoms, complications, electrocardiogram and 24-hour dynamic electrocardiogram.

ELIGIBILITY:
Inclusion Criteria:

* Persistent AF is defined as AF that persists without interruption for 7 days (electrocardiogram data or Holter), atrial fibrillation cannot be prevented in patients who orally take class I and III antiarrhythmic drugs, and patient age is <80 years.

Exclusion Criteria:

* •left ventricular dysfunction

  * atrial thrombosis
  * valvular heart disease
  * hyperthyroidism
  * patients who underwent prosthetic heart valve replacement
  * patients with previous history of atrial fibrillation ablation
  * pregnant women
  * patients with existing liver and kidney disease
  * malignant tumors
  * hematological system diseases
  * patients who underwent prosthetic heart valve replacement

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2018-08-28 (Actual); Primary Completion 2020-11-28 (Actual); Study Completion 2020-12-28 (Actual)

PRIMARY OUTCOMES:
Left atrial function of postoperative | 1-12 month
  Transthoracic echocardiography
Atrial electrical activity | During the operation
  Electrophysiological examination

SECONDARY OUTCOMES:
C-Reactive Protein | 1-12 month
  Blood samples are extracted in all patients to detected
leukocyte assessed | 1-12 month
  Blood samples are extracted in all patients to detected
Neutrophil assessed | 1-12 month
  Blood samples are extracted in all patients to detected
Lymphocyte assessed | 1-12 month
  Blood samples are extracted in all patients to detected
Neutrophil/Lymphocyte | 1-12 month
  Blood samples are extracted in all patients to detected
B type natriuretic peptide assessed | 1-12 month
  Blood samples are extracted in all patients to detected
Coagulation index assessed | 1-6 month
  Blood samples are extracted in all patients to detected
Change of P wave | 1-12 month
  Electrocardiogram
homocysteine assessed | 1-12 month
  Blood samples are extracted in all patients to detected
β2-microglobulin assessed | 1-12 month
  Blood samples are extracted in all patients to detected

CONTACTS AND LOCATIONS:
Locations (1):
- Second Hospital of Hebei Medical University, Shijiazhuang, Hebei, China